CLINICAL TRIAL: NCT06456567
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Telitacicept Compared to Placebo in Patients With Moderately to Severely Active Systemic Lupus Erythematosus (REMESLE-2)
Brief Title: A Study of Telitacicept for the Treatment of Moderately to Severely Active Systemic Lupus Erythematosus (REMESLE-2)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor business decision
Sponsor: Vor Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC18G002
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental): Telitacicept + Standard of Care (SOC)
  Interventions: Biological: Telitacicept
- Placebo (Placebo Comparator): Placebo + Standard of Care (SOC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept — Subcutaneous injection
  Arms: Telitacicept
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of telitacicept in the treatment of moderately to severely active SLE.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune disease with heterogeneous manifestations and disease course. Despite advances in medical care, there are still significant unmet needs in SLE with diminished health-related quality of life (HRQoL), persistent disease activity, disease flares, intolerance to standard of care (SOC) therapies, and development of organ damage and co-morbidities.

Telitacicept is a fully human TACI-Fc fusion protein that targets B lymphocyte stimulator (BLyS) and a proliferating-inducing ligand (APRIL). Blocking the interaction of BLyS and APRIL with their cell membrane receptors (TACI, B-cell maturation antigen (BCMA), and B-cell activating factor receptor (BAFF-R) would inhibit B cell proliferation and maturation, suppresses immune responses and may alleviate autoimmune symptoms.

This is a multicenter, randomized, double-blind, placebo-controlled, phase 3 study to evaluate the efficacy and safety of telitacicept added to standard of care (SoC) therapy compared to placebo with SoC therapy in subjects with moderately to severely active SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-70 years at screening.
2. Has a diagnosis of SLE for at least 6 months prior to the screening visit.
3. Meets the 2019 EULAR/ACR Classification criteria for SLE.
4. Moderately to severely active SLE definined by the following:

   1. SELENA SLEDAI total score ≥6 points with clinical SLEDAI score ≥4 points at screening;
   2. BILAG organ system scores of at least 1A or 2B at screening.
5. Clinical SLEDAI score of ≥4 at Day 0 prior to randomization.
6. At least one positive serologic parameter within the screening period.
7. Currently receiving at least one of the SOC SLE medications: oral corticosteroid, antimalarial and/or immunosuppressive agent.

Exclusion Criteria:

1. Active lupus nephritis undergoing induction therapy or unstable renal diseases within 12 weeks prior to screening.
2. Active or unstable neuropsychiatric SLE.
3. Autoimmune or rheumatic disease other than SLE.
4. History of arterial or venous thromboembolism or microangiopathy within 12 months prior to screening.
5. History of non-SLE disease requiring treatment with oral or parenteral. glucocorticosteroids for more than a total of 2 weeks within the last 24 weeks prior to screening.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
SLE Responder Index (SRI-4) | Week 52
  Proportion of subjects achieving an SLE Responder Index (SRI-4) response

SECONDARY OUTCOMES:
SLE Responder Index (SRI-4) | Week 24
  Proportion of subjects achieving an SLE Responder Index (SRI-4) response
Achieve and sustain a low dose of corticosteriods | Week 52
  Proportion of subjects achieving the target of corticosteroids reduction.
SLE Responder Index (SRI-4) and sustaining a low dose of corticosteriods | Week 52
  Proportion of patients achieving an SRI-4 response at Week 52, while achieving and maintaining corticosteroids reduction.
BILAG-based Combined Lupus Assessment (BICLA) Response | Week 52
  Proportion of patients achieving a BILAG-based Combined Lupus Assessment (BICLA) response at Week 52
Time to Flare | Up to Week 52
  Time to flare assessed by SELENA-SLEDAI Flare Index (SFI) from baseline through Week 52
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Week 52
  Proportion of patients achieving clinically meaningful improvement in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at Week 52

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hemet site, Hemet, California
  - Menifee site, Menifee, California
  - Rockford site, Rockford, Illinois
  - Stafford site, Stafford, Texas

IPD SHARING:
Plan to Share IPD: No